CLINICAL TRIAL: NCT03639155
Title: A Randomized, Open-Label, Single-Dose, Two-Period Crossover Study in Healthy Adults to Assess Bioequivalence Between Test and Reference Formulations of Vadadustat 150 mg Tablets
Brief Title: A Study in Evaluating Bioequivalence Between Test and Reference Formulations of Vadadustat Tablets in Healthy Adults
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Akebia Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: AKB-6548-CI-0027
Record Dates: First submitted 2018-06-12; First posted 2018-08-21 (Actual); Last update posted 2019-03-22 (Actual); Status verified 2019-03

CONDITIONS: Healthy
Keywords: vadadustat; AKB-6548; hypoxia-inducible factor; HIF; hypoxia-inducible factor prolyl-hydroxylase inhibitor; HIF-PHI
MeSH Terms: interventions — vadadustat

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Regimen A (Experimental): vadadustat reference tablets
  Interventions: Drug: vadadustat reference tablets
- Regimen B (Experimental): vadadustat test tablets
  Interventions: Drug: vadadustat test tablets

INTERVENTIONS:
Drug: vadadustat reference tablets — oral tablet
  Other Names: AKB-6548
  Arms: Regimen A
Drug: vadadustat test tablets — oral tablet
  Other Names: AKB-6548
  Arms: Regimen B

SUMMARY:
This study is to assess the bioequivalence of a test formulation of vadadustat (A) compared to a reference formulation of vadadustat (B)

DETAILED DESCRIPTION:
This is a randomized, open-label, single-dose, two-period crossover study in healthy adults to assess the bioequivalence of a test formulation of vadadustat compared to the reference formulation of vadadustat. Blood samples for vadadustat PK will be collected at pre-dose (0 hour) and at 0.5, 1, 1.5, 2, 3, 4, 6, 9, 12, 18, 24, 32, 40, and 48 hours post-dose.

ELIGIBILITY:
Inclusion Criteria:

* Between 18 and 55 years of age, inclusive, at time of informed consent.
* Healthy subjects per Investigator judgment as documented by the medical history, physical examination, vital sign assessments, 12-lead electrocardiogram (ECG), clinical laboratory assessments, and general observations.
* Minimum weight of 45 kg with Body mass index (BMI) between 18 and 29.5 kg/m2, inclusive.
* Understands the procedures and requirements of the study and provides written informed consent and authorization for protected health information disclosure
* Willing and able to comply with the requirements of the study protocol.

Exclusion Criteria:

* Current or past history of cardiovascular, cerebrovascular, pulmonary, gastrointestinal, hematologic, renal, hepatic, immunologic, metabolic, urologic, neurologic, dermatologic, psychiatric, or other major disease, history of cancer (except non-melanoma skin cancer) or history of chemotherapy use.
* Any surgical or medical condition or history that may potentially alter the absorption, metabolism, or excretion of study treatment, such as, but not limited to gastric bypass surgery or gastric or duodenal ulcers.
* History of severe allergic or anaphylactic reactions.
* Chronic daily medication use.
* History of drug abuse
* Excessive alcohol consumption
* Smoking and the use of nicotine-containing products
* Consumption of grapefruit or grapefruit juice, pomelo, star fruit, Seville or Moro (blood) orange, or their associated products
* Participation in another clinical trial or exposure to any investigational agent.
* Donation of blood or significant blood loss or plasma donation.
* Any condition that would interfere with the ability to provide informed consent, comply with study instructions, or which might confound the interpretation of the study results or put the patient at undue risk.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 50 (Actual)
Dates: Start 2018-04-12 (Actual); Primary Completion 2018-05-23 (Actual); Study Completion 2018-05-23 (Actual)

PRIMARY OUTCOMES:
Area under plasma concentration-time curve from 0 to last quantifiable concentration (AUClast) | Baseline visit, 48 hours
Area under plasma concentration-time curve from 0 to infinity (AUCinf) | Baseline visit, 48 hours
Area under plasma concentration-time curve from 0 to last sampling point (AUCall) | Baseline visit, 48 hours
Observed maximum concentration (Cmax) | Baseline visit, 48 hours

SECONDARY OUTCOMES:
Time to reach Cmax | Baseline visit, 48 hours
Time to reach Tmax | Baseline visit, 48 hours
Mean residence time (MRT) | Baseline visit, 48 hours
Elimination rate constant (Kel) | Baseline visit, 48 hours
Apparent total body clearance (CL/F) | Baseline visit, 48 hours
Apparent volume of distribution (Vd/F) | Baseline visit, 48 hours
Terminal half-life (t1/2) | Baseline visit, 48 hours

CONTACTS AND LOCATIONS:
Overall Officials: Akebia, Study Director — Sponsor GmbH
Locations (1):
- Research Site, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: Undecided